CLINICAL TRIAL: NCT04377282
Title: The Effect of Buckwheat on Blood Glucose, Satiety and Food Intake
Brief Title: The Effect of Buckwheat and Couscous on Satiety and Food Intake in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Saint Vincent University (Other)
Responsible Party: Principal Investigator, Bohdan Luhovyy, Associate Professor, Mount Saint Vincent University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-085
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Food; Eating; Appetite

STUDY DESIGN:
Intervention Model Description: Randomized crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Buckwheat (Experimental): Cooked buckwheat
  Interventions: Other: Food-1
- Couscous (Experimental): Cooked couscous
  Interventions: Other: Food-2
- Water (Experimental): Potable water
  Interventions: Other: Food-3

INTERVENTIONS:
Other: Food-1 — Cooked buckwheat
  Arms: Buckwheat
Other: Food-2 — Cooked couscous
  Arms: Couscous
Other: Food-3 — Water
  Arms: Water

SUMMARY:
A diet rich in whole grains has been linked to multiple beneficial health outcomes, including cardiovascular health, weight loss and a decreased risk of acquiring type 2 diabetes. However, grain products vary due to their botanical origin, composition, and post-harvest processing. While wheat is considered a dominant grain crop in Canada, the minor crops, including gluten-free buckwheat, become popular alternatives to wheat products such as couscous. Both buckwheat groats and couscous are traditionally consumed in the form of the porridge or side dish, however, their acute effects on satiety and food intake remain unknown. The objective of this study is to investigate the short-term effects of couscous and buckwheat on satiety and short-term food intake in young adult males.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 18-30 years

Exclusion Criteria:

* Smokers
* Taking medication
* Breakfast skippers

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Food intake | 120 minutes
  The amount of energy (kcal) consumed ad libitum with the test meal (pizza lunch) two hours later.
Subjective appetite | 0-120 minutes
  The subjective assessment of appetite parameters including a desire to eat, fullness, hunger and a prospective food consumption measured with 100 mm Visual Analogue Scales with two opposite statements at each end (e.g., for the hunger scale, 0 mm means not hungry at all, and 100 mm means very hungry).

SECONDARY OUTCOMES:
Subjective feeling of physical comfort | 0-120 minutes
  The subjective assessment of wellness and gastrointestinal symptoms including a feeling of nausea, diarrhea, flatulence, and other parameters measured with 100 mm Visual Analogue Scales with two opposite statements at each end.
Subjective perception of food palatability (pleasantness) | 0, 120 minutes
  The pleasantness of the meals measured with 100 mm Visual Analogue Scales with two opposite statements at each end (e.g., 0 mm means that food is not pleasant at all, and 100 mm means that the food is very pleasant).

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan L. L Luhovyy, PhD, Principal Investigator — Mount Saint Vincent University
Locations (1):
- Mount Saint Vincent University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No